CLINICAL TRIAL: NCT00567931
Title: A Phase 1 Study of 1-Methyl-D-tryptophan in Patients With Advanced Malignancies
Brief Title: 1-Methyl-D-Tryptophan in Treating Patients With Metastatic or Refractory Solid Tumors That Cannot Be Removed By Surgery
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00268; NCI-2009-00268 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); MCC-FL065; CDR0000576700; MCC 15267 (Other: H. Lee Moffitt Cancer Center and Research Institute); 8045 (Other: CTEP); N01CM00100 (NIH); P30CA076292 (NIH); NCT00617422 (obsolete NCT alias)
Record Dates: First submitted 2007-12-04; First posted 2007-12-05 (Estimated); Last update posted 2014-07-24 (Estimated); Status verified 2014-07

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
MeSH Terms: interventions — 1-methyltryptophan

ARMS (1):
- Treatment (Immunomodulating therapy) (Experimental): Patients receive oral 1-methyl-d-tryptophan (1-MT) once or twice daily on days 1-28. Treatment repeats every 28 days for up to 12 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: 1-methyl-d-tryptophan; Other: pharmacological study; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: 1-methyl-d-tryptophan — Given orally
  Other Names: indoximod
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase I trial is studying the side effects and best dose of 1-methyl-D-tryptophan in treating patients with metastatic or refractory solid tumors that cannot be removed by surgery. Biological therapies, such as 1-methyl-D-tryptophan, may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth and by stimulating the immune system.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the toxicity, safety, and pharmacokinetics of escalating doses of 1-methyl-d-tryptophan (1-MT), a competitive inhibitor of the enzyme indoleamine 2, 3-dioxygenase (IDO), in patients with advanced malignancies.

II. To establish a maximally tolerated dose (MTD) or maximally biological effective dose (MBED) of 1-MT for future phase II and III trials.

SECONDARY OBJECTIVES:

I. To assess the ratio of kynurenine to tryptophan in patient blood samples as a means of assessing the effect of 1MT on in vivo IDO activity.

II. To ascertain the ability of 1-MT to decrease the number of T-regulatory cells thereby allowing the immune system to target tumor antigens more effectively.

III. To analyze the IDO expression of different tumor types through IDO immunohistochemical staining of paraffin-preserved specimens.

IV. To perform high performance liquid chromatography on patient urine samples to assess how 1-MT is cleared renally.

OUTLINE: This is a dose-escalation study.

Patients receive oral 1-methyl-d-tryptophan (1-MT) once or twice daily on days 1-28. Treatment repeats every 28 days for up to 12 courses in the absence of disease progression or unacceptable toxicity.

Blood and urine samples are assessed to characterize the pharmacokinetics of 1-MT and renal clearance rate by high performance liquid chromatography, measure tryptophan and kynurenine levels by functional assays, and measure the response of regulatory CD4+ CD25+ T cells by intracellular staining and flow cytometry. Paraffin-embedded tissue samples are analyzed for indoleamine 2, 3-dioxygenase (IDO) expression by immunohistochemical staining.

After completion of study treatment, patients are followed up for 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed solid malignancy that is metastatic or unresectable and for which standard effective antineoplastic therapy does not exist or is no longer effective
* Patients are eligible for enrollment into the trial regardless of the types of previous therapies administered
* Patients with known brain metastases will only be eligible after their tumors have been treated with definitive resection and/or radiotherapy and they are neurologically stable for at least 1 month off steroids

  * No known untreated brain metastases
* ECOG performance status (PS) 0-2 OR Karnofsky PS 60-100%
* Life expectancy > 4 months
* WBC ≥ 3,000/μL
* ANC ≥ 1,500/μL
* Platelet count ≥ 100,000/μL
* Total bilirubin ≤ 1.5 times upper limit of normal (ULN)
* AST and ALT ≤ 2.5 times ULN
* Creatinine normal OR creatinine clearance ≥ 60 mL/min
* No history of gastrointestinal disease causing malabsorption or obstruction, including, but not limited to, any of the following:

  * Crohn's disease
  * Celiac sprue
  * Tropical sprue
  * Bacterial overgrowth/blind-loop syndrome
  * Strictures
  * Adhesions
  * Achalasia
  * Bowel obstruction
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective double-method contraception during and for at least 1 month after completion of study treatment
* No history of allergic reactions (significant urticaria, angioedema, anaphylaxis) attributed to compounds of similar chemical or biologic composition to 1-methyl-d-tryptophan (including L-tryptophan or 5-hydroxy-tryptophan supplements)
* No active autoimmune disease (i.e., psoriasis, extensive atopic dermatitis, asthma, inflammatory bowel disorder, multiple sclerosis, uveitis, vasculitis), chronic inflammatory condition, or any condition requiring concurrent use of any systemic immunosuppressants or steroids for any reason
* Mild-intermittent asthma requiring only occasional beta-agonist inhaler use or mild localized eczema allowed
* No uncontrolled concurrent illness including, but not limited to, any of the following:

  * Ongoing or active infection
  * Symptomatic congestive heart failure
  * Unstable angina pectoris
  * Myocardial infarction or percutaneous coronary interventions within the past 6 months
  * Cardiac arrhythmia
  * Active autoimmune diseases
  * Major psychiatric illness or social situation that would limit compliance with study requirements as judged by the primary investigator at each site
* Patients with well-controlled, chronic medical conditions under the supervision of the patient's primary physician (i.e., hypertension, hyperlipidemia, coronary heart disease, diabetes mellitus) are eligible
* No HIV-positive patients or patients with other acquired/inherited immunodeficiencies
* No other active malignancy
* No concurrent immunosuppressants, including steroids
* Recovered from all prior therapy
* No prior gastric bypass surgery
* No prior extensive small bowel resection
* No prior experimental active immunotherapy consisting of targeted monoclonal antibodies or pharmaceutical compounds

  * Commercially available active immunotherapy (e.g., adjuvant interferon) must have completed therapy over 1 year prior to enrollment and have no evidence of autoimmune sequelae
* Prior therapy with approved monoclonal antibodies (e.g., bevacizumab, cetuximab, panitumumab, or trastuzumab) allowed
* At least 4 weeks since prior and no other concurrent investigational agents
* More than 4 weeks since prior chemotherapy or radiotherapy (6 weeks for nitrosoureas or mitomycin C)
* No concurrent supplements containing L-tryptophan or derivatives
* No patients with an allo-transplant of any kind (including those with a xenograft heart valve)
* No other concurrent commercial agents or therapies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2007-10; Primary Completion 2012-07 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events, graded according to the standard Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 | Up to 4 weeks
  All patients who receive any amount of the study drug will be evaluable for toxicity.
MTD or MBED of 1-Methyl-D-tryptophan | Up to 4 weeks
  A dose limiting toxicity (DLT) will be defined as any adverse events (AEs) occurring during any course when considered possibly, probably, or definitely related to therapy that is part of this study. Unacceptable AEs including any grade 3 or greater toxicity possibly, probably, or definitely due to the study drug (except oral intolerance). The MBED will be determined retrospectively after all data has been collected and an MTD has been determined.

SECONDARY OUTCOMES:
Pharmacokinetics of 1-methy-D-tryptophan | At 0, 0.5, 1, 2, 4, 6, 8, 12, 24, and 48 hours after administration
  Analyses of secondary endpoints will mainly be of exploratory nature. If needed, non-parametric methods such as the signed rank test and/or Spearman correlation coefficient will be considered to explore preliminarily the treatment effect on the secondary endpoints and its relationships with various potential biomarkers and therapeutic targets.
Change in the tryptophan kynurenine ratio | Baseline to up to week 5
  Descriptive statistics such as means, medians, interquartiles, and standard deviations (SDs) or frequencies and percentages will be reported. When appropriate, confidence intervals also will be included. Change data contrasting post-treatment vs baseline will be summarized similarly. If needed, non-parametric methods such as the signed rank test and/or Spearman correlation coefficient will be considered to explore preliminarily the treatment effect on the secondary endpoints and its relationships with various potential biomarkers and therapeutic targets.
Change in the number of circulating CD4+ CD25+ Treg cells | Baseline to up to 4 weeks after completion of study treatment
  Descriptive statistics such as means, medians, interquartiles, and SDs or frequencies and percentages will be reported. When appropriate, confidence intervals also will be included. Change data contrasting post-treatment vs baseline will be summarized similarly. If needed, non-parametric methods such as the signed rank test and/or Spearman correlation coefficient will be considered to explore preliminarily the treatment effect on the secondary endpoints and its relationships with various potential biomarkers and therapeutic targets.
IDO expression in tumor tissue | At baseline
  Descriptive statistics such as means, medians, interquartiles, and SDs or frequencies and percentages will be reported. When appropriate, confidence intervals also will be included. Change data contrasting post-treatment vs baseline will be summarized similarly. If needed, non-parametric methods such as the signed rank test and/or Spearman correlation coefficient will be considered to explore preliminarily the treatment effect on the secondary endpoints and its relationships with various potential biomarkers and therapeutic targets.

CONTACTS AND LOCATIONS:
Overall Officials: Scott Antonia, Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (2):
- United States (2):
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Virginia Commonwealth University, Richmond, Virginia